CLINICAL TRIAL: NCT06148480
Title: Perinatal Transmission of Multi-drug Resistant (MDR) Bacteria
Brief Title: Perinatal Transmission of MDR Bacteria
Acronym: ACQUIRE
Status: Recruiting | Type: Observational
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Mehreen Arshad, Assistant Professor of Pediatrics, Ann & Robert H Lurie Children's Hospital of Chicago
Other Study IDs: IRB 2020-3331
Record Dates: First submitted 2023-11-20; First posted 2023-11-28 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: E. Coli Infection; Multi-antibiotic Resistance
MeSH Terms: conditions — Escherichia coli Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Mothers will be asked to self-collect perineal (x2) and rectal swabs (x2) while they are admitted in the hospital. Infant stool samples will be collected between the first 24-48 hrs. of life. We will also be collecting infant stool samples at day 7 of life (+/- 2 days).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mother-Infant Dyads: Women and their neonates admitted to the postpartum floor will be enrolled after being screened for the exclusion criteria

SUMMARY:
The investigators aim to conduct a prospective surveillance study of mothers and their infants born vaginally or by scheduled C-section and who are admitted to Northwestern Medicine Prentice Women's Hospital to determine the prevalence of ESBL-E carriage in healthy post-partum women and the transmission rate of these strains to their infants. Using whole genome sequencing and a comparative genomics approach the investigators will determine the relatedness of strains among mother-infant dyads as well as identify genetic regions common to transmitted strains. It is hypothesize that; 1) given the diverse population of Chicago there will be a significant rate of gut colonization with ESBL-E among mothers admitted to Prentice, 2) ESBL-E strains isolated from neonates will be identical to those from their mothers and 3) genetic determinants of transmission are conserved across ESBL E. coli strains that are perinatally transmitted. These hypotheses will be tested using the following Aims:

Aim 1: Determine the prevalence of ESBL-E gut colonization and rate of perinatal transmission among mother-infant dyads Aim 2: Identify genetic determinants of transmission common to ESBL E. coli that are perinatally transmitted.

The long-term goal is to understand the unique features of persistent gut and vaginal ESBL-E colonizers and identify genetic and molecular elements that could be attractive therapeutic targets to decrease the burden of ESBL-E colonization and perinatal transmission.

DETAILED DESCRIPTION:
The rapid rise of multi-drug resistant Enterobacteriaceae (MDR-E) is severely threatening the way we treat common infectious diseases. A particularly vulnerable population are neonates where a delay in the treatment of MDR-E sepsis can be fatal. Additionally, highly drug resistant bacteria such as the pandemic E. coli ST131 strain are persistent gut and vaginal colonizers (1). In animal models of gut colonization, these strains out-compete drug-sensitive, commensal Escherichia coli. Early life exposure to MDR-E could, therefore, have long-lasting effects on the developing microbiome and overall child health (2).

Among extra-intestinal pathogenic Enterobacteriaceae, resistance against a number of antibiotics, especially the beta-lactams, has rapidly risen in the last decade. Since the gut is a major reservoir of these pathogens even in otherwise healthy individuals it is likely that there is a concomitant increase in gut colonization with extended spectrum beta-lactamase producing Enterobacteriaceae (ESBL-E) among the general population (3, 4). Even in regions with a low prevalence of community acquired ESBL-E infections, perinatal transmission occurs in 35% of infants born to mothers colonized with these strains (5). It has recently been shown that healthy infants in South Asia, a region with a high use of antibiotics per capita, are carriers of ESBL-E (6). In vitro studies suggest that ESBL E. coli isolated from these infants have a higher growth potential than commensal E. coli. Using a murine model of perinatal transmission of E. coli, it was shown that some of the ESBL E. coli strains adept in human infant gut colonization can also readily colonize pregnant dams and be perinatally transmitted. The burden of ESBL-E colonization among pregnant women and their neonates in the US and the genetic determinants of perinatal transmission are unknown.

The investigators aim to conduct a prospective surveillance study of mothers and their infants born vaginally and who are admitted to Northwestern Medicine Prentice Women's Hospital to determine the prevalence of ESBL-E carriage in healthy post-partum women and the transmission rate of these strains to their infants. Using whole genome sequencing and a comparative genomics approach they will determine the relatedness of strains among mother-infant dyads as well as identify genetic regions common to transmitted strains. It is hypothesized that; 1) given the diverse population of Chicago there will be a significant rate of gut colonization with ESBL-E among mothers admitted to Prentice, 2) ESBL-E strains isolated from neonates will be identical to those from their mothers and 3) genetic determinants of transmission are conserved across ESBL E. coli strains that are perinatally transmitted. These hypotheses will be tested using the following Aims:

Aim 1: Determine the prevalence of ESBL-E gut colonization and rate of perinatal transmission among mother-infant dyads Aim 2: Identify genetic determinants of transmission common to ESBL E. coli that are perinatally transmitted.

The long-term goal is to understand the unique features of persistent gut and vaginal ESBL-E colonizers and identify genetic and molecular elements that could be attractive therapeutic targets to decrease the burden of ESBL-E colonization and perinatal transmission.

ELIGIBILITY:
Inclusion Criteria:

* Women that are admitted to Northwestern Medicine Women's Hospital that have delivered an infant vaginally or have had a scheduled C-section without preceding labor.
* Infants that are born vaginally who are healthy and do not require transfer to the NICU for any reason.

Exclusion Criteria:

* Temperature >38 Celsius in labor
* Caesarean section after labor
* Rupture of membranes or done emergently
* Antibiotic use in last trimester including for GBS+
* Delivery at <35 weeks
* Immunocompromised host including being HIV+
* Infant requiring transfer to NICU for any reason and infants who are transferred to the NICU.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Mothers and their infants born vaginally or by scheduled c-section and who are admitted to Northwestern Medicine Prentice Women's Hospital
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-07-17 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
ESBL-E Prevalence | Baseline
  Determine the proportion of women in the post-partum period that are colonized with ESBL-E
Transmission Among Mother-Infant Dyads | Baseline
  Determine the proportion of neonates that acquire ESBL-E strains perinatally
Persistence of ESBL-E Colonization | 7 days from baseline
  For determine colonization of ESBL-E organisms in neonates 7 days after birth.

SECONDARY OUTCOMES:
Genetic Determinants of ESBL-E | Baseline
  Identifying specific genes that are important for successful perinatal transmission of ESBL-E

CONTACTS AND LOCATIONS:
Overall Officials: Mehree Arshad, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Prentice Women's Hospital, Chicago, Illinois, United States